CLINICAL TRIAL: NCT01261494
Title: A Pilot Study to Evaluate the Efficacy and Safety of GFT505 (80mg) Orally Administered Once Daily for 12 Weeks in Patients With Type 2 Diabetes Mellitus. A Multicentre, Randomised, Double Blind, Placebo-Controlled Study.
Brief Title: Study With GFT505 (80mg) Versus Placebo in Patients With Type 2 Diabetes Mellitus
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Genfit (Industry)
Responsible Party: Product Development Department, Genfit
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: GFT505-210-5; 2010-021986-60 (EudraCT Number)
Record Dates: First submitted 2010-12-13; First posted 2010-12-16 (Estimated); Last update posted 2011-07-13 (Estimated); Status verified 2011-07

CONDITIONS: Type II Diabetes Mellitus
Keywords: Diabetes Mellitus, Type 2; Glucose Metabolism Disorders; Metabolic Diseases; Cardiovascular Diseases; PPARs; OGTT
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Glucose Metabolism Disorders; Metabolic Diseases; Cardiovascular Diseases | interventions — 2-(2,6-dimethyl-4-(3-(4-(methylthio)phenyl)-3-oxo-1-propenyl)phenoxyl)-2-methylpropanoic acid

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- GFT505 80mg (Experimental)
  Interventions: Drug: GFT505 80mg
- Matching placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: GFT505 80mg — hard gelatin capsules dosed at 20mg,oral administration,4 capsules per day before breakfast
  Arms: GFT505 80mg
Drug: Placebo — hard gelatin capsules,oral administration,4 capsules per day before breakfast
  Arms: Matching placebo

SUMMARY:
This study is expected to demonstrate the anti-diabetic efficacy of 3-months treatment with GFT505 (80 mg/d) on Glycosylated Haemoglobin A1c (HbA1C) and fasting plasma glucose.

And to assess the tolerability and safety of once-a-day administrations of oral doses of GFT505 for 12 weeks in patients with type 2 diabetes mellitus.

DETAILED DESCRIPTION:
The study period per patient is 16-20 weeks maximum and is conducted as follows :

* Run-in period: 2 weeks or 6 weeks for patients under fibrate treatment at screening (4 weeks fibrate wash-out + 2 weeks placebo run-in);
* Treatment period: 12 weeks;
* Follow-up period: 2 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Male or post-menopausal female (defined as >12 months since last menstrual period) or surgical menopause. If hormonal replacement therapy, it should be stable at least for 6 months prior to screening.
* Body Mass Index ≥27 and ≤45 kg/m².
* Drug-Naive patients with type 2 diabetes mellitus (non insulin dependent diabetes). Patients should not be treated by insulin or other diabetes medication for the last 3 months prior to screening. Patients treated for less than 4 weeks with insulin may be included in the study.
* HbA1c ≥ 7.0% and <9.5%.
* Antibody glutamate decarboxylase acid (Anti-GAD) negative for patients aged less than 40 years.

Exclusion Criteria:

* Type I Diabetes Mellitus.
* Blood Pressure > 160 / 95 mmHg.
* Lipid-lowering drugs such as fibrates.
* Fasting Plasma Glucose (FPG) ≥ 240 mg/dL.
* Triglycerides (TG) > 400 mg/dL.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 97 (Actual)
Dates: Start 2010-12; Primary Completion 2011-06 (Actual); Study Completion 2011-06 (Actual)

PRIMARY OUTCOMES:
HbA1c | 12 weeks
  To evaluate after 12 weeks of oral administration of double blind treatment the change from baseline in HbA1c level achieved with GFT505 80mg versus placebo. Evaluation will be made during the selection period, prior any drug intake, and 4, 8, 12 weeks after the first treatment intake as well as 2 weeks after the last treatment intake (follow up period).

SECONDARY OUTCOMES:
Oral Glucose Tolerance Test (OGTT) | 12 weeks
  To evaluate the changes from baseline to end of treatment in OGTT parameters. Evaluation will be made prior the first treatment intake and 12 weeks after the first treatment intake.
Fasting Plasma Glucose | 12 weeks
  To evaluate the changes from baseline to end of treatment in fasting plasma Glucose. Evaluation will be made during the selection period, prior any drug intake, and 4, 8, 12 weeks after the first treatment intake as well as 2 weeks after the last treatment intake (follow up period).
Insulin resistance Index [fasting insulin and homeostasis model assessment of insulin resistance (HOMA-IR)] | 12 weeks
  To evaluate the changes from baseline to end of treatment in insulin resistance index. Evaluation will be made during the selection period, prior any drug intake, and 4, 8, 12 weeks after the first treatment intake as well as 2 weeks after the last treatment intake (follow up period).

CONTACTS AND LOCATIONS:
Overall Officials: Rémy HANF, Development Director, Study Director — Genfit, France; Bertrand CARIOU, Pr., Study Chair — University Hospital of Nantes, France
Locations (28):
- Bosnia and Herzegovina (2):
  - Site n°12, Banja Luka
  - Site n°11, Sarajevo
- Latvia (3):
  - Site n°22, Riga
  - Site n°21, Riga
  - Site n°23, Valmiera
- Moldova (3):
  - Site n°41, Bălţi
  - Site n°42, Chisinau
  - Site n°43, Chisinau
- North Macedonia (3):
  - Site n°33, Bitola
  - Site n°31, Skopje
  - Site n°32, Skopje
- Romania (12):
  - Site n°72, Oradea, Bihor County
  - Site n°66, Buzău, Buzău
  - Site n°64, Cluj-Napoca, Cluj
  - Site n°65, Baia Mare, Maramureş
  - Site n°63, Târgu Mureş, Mureș County
  - Site n°62, Târgu Mureş, Mureș County
  - Site n°71, Ploieşti, Prahova
  - Site n°70, Ploieşti, Prahova
  - Site n°61, Sibiu, Sibiu County
  - Site n°67, Bucharest
  - Site n°69, Bucharest
  - Site n°68, Bucharest
- Serbia (5):
  - Site n°52, Belgrade
  - Site n°53, Belgrade
  - Site n°56, Belgrade
  - Site n°54, Kragujevac
  - Site n°51, Niš